CLINICAL TRIAL: NCT01811446
Title: Evaluation of Muscle Stimulation Efficiency in Challenging Subjects: A Pilot Study
Brief Title: Evaluation of Muscle Activation Efficiency in Challenging Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Niveus Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP-2.00
Record Dates: First submitted 2013-03-12; First posted 2013-03-14 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Obesity; COPD
MeSH Terms: conditions — Obesity; Pulmonary Disease, Chronic Obstructive

ARMS (2):
- Obese (Experimental): Subjects with BMI > 30
  Interventions: Device: Muscle Activation with Niveus and Intelect Devices
- COPD (Experimental): Non-hospitalized COPD patients
  Interventions: Device: Muscle Activation with Niveus and Intelect Devices

INTERVENTIONS:
Device: Muscle Activation with Niveus and Intelect Devices — Subjects will receive muscle activation technology from the Niveus device on one leg and from the Intelect (commercially-available third-party) device on the other. The order of use and the leg applied to will be randomized.

SUMMARY:
The purpose of this study is to determine whether muscle activation can be accomplished more effectively and comfortably in challenging subjects using novel configurations of an activation device. A novel device will be compared side by side with a market leading device.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30 (Wing 1 of study)
* Non-hospitalized with confirmed diagnosis of COPD (Wing 2 of study)

Exclusion Criteria:

* Age < 18 years
* Subject has an implanted pacemaker/defibrillator
* Subject diagnosed with epilepsy
* Subject has implanted metallic femoral rods
* Subject is chair- or bed-bound
* Subject has neuromuscular disease or abnormalities
* Subject BMI > 45
* Evidence of disease or condition that, in the opinion of the investigator, may compromise the conduct of or results of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-03; Primary Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Intensity Required | During treatment
  Intensity required to achieve target levels of muscle contraction

SECONDARY OUTCOMES:
Comfort | During treatment
  Comfort of stimulation will be assessed at various intensity levels using a widely-used discomfort scale

CONTACTS AND LOCATIONS:
Overall Officials: Bahman Nouri, MD, Principal Investigator — El Camino Hospital
Locations (1):
- Fogarty Clinical Research, Mountain View, California, United States